CLINICAL TRIAL: NCT04925219
Title: Remotely Supervised Exercise Versus Self-Directed Exercise: Phase II Safety and Efficacy Study
Brief Title: REmotely Supervised Exercise Therapy Trial 2
Acronym: RESET2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2987694
Record Dates: First submitted 2021-03-24; First posted 2021-06-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Claudication, Intermittent; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Pilot 2 arm RCT
Who Masked: Outcomes Assessor
Masking Description: Independent assessment of absolute walking distance and QoL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remotely supervised exercise (Experimental): Best medical therapy including aspirin 75mg od + rivaroxaban 2.5mg bd (if not tolerated clopidogrel 75mg od), atorvastatin 80mg and smoking cessation referral as per NICE guideline for PAD.
  Intervention = electronic walking log and fortnightly video/telephone call with physiotherapist for 3 months.
  Interventions: Behavioral: Remotely supervised exercise programme
- Self-directed exercise (Active Comparator): Best medical therapy including aspirin 75mg od + rivaroxaban 2.5mg bd (if not tolerated clopidogrel 75mg od), atorvastatin 80mg and smoking cessation referral as per NICE guideline for PAD.
  Control = electronic walking log and instructions to exercise 4 times per week for 3 months
  Interventions: Behavioral: Self-directed exercise

INTERVENTIONS:
Behavioral: Remotely supervised exercise programme — Electronic walking log Fortnightly video/telephone calls with physiotherapist
  Arms: Remotely supervised exercise
Behavioral: Self-directed exercise — Electronic walking log and instructions to exercise 4 times per week.
  Arms: Self-directed exercise

SUMMARY:
Supervised exercise for intermittent claudication is a first line therapy for peripheral arterial disease, as recommended by the National Institute for Health and Clinical Excellence and the European Society for Vascular Surgery. However 2/3 of British trusts cannot implement this due to gym availability, costs, travel time and the requirement for social distancing.

During the COVID-19 lockdown the investigators successfully performed a feasibility study for remotely supervised exercise using an electronic walking log and fortnightly video calls with a physiotherapist.

RESET2 aims to compare the benefits of and adherence to remotely supervised exercise with self-directed exercise to absolute walking distance.

DETAILED DESCRIPTION:
Design A single centre, pilot, randomised controlled trial at Mid and South Essex Hospitals Foundation Trust. The study is unfunded and sponsored by Mid and South Essex Hospitals National Health Service Trust.

Sample size This is a pilot randomised controlled trial to generate a sample size calculation for a larger trial.

Based on the feasibility data from RESET1 and the published results of supervised exercise, the expected benefit of remotely supervised exercise is about 180 metres extra walking distance, with a standard deviation of 150m in both groups.

With alpha=0.05 (5% false positive rate) and beta=0.1 (90% power), 16 patients in each arm are required to demonstrate a mean difference in the primary endpoint of 180 metres, using a 2 sided t-test (MedCalc statistical software, Belgium).

The sample size will be 20+20 patients from Mid and South Essex Trust vascular outpatient clinics.

Follow up There will be 3 assessment visits: baseline, 3 months and 6 months performed with a study clinician.

The primary endpoint will be measured blind to treatment allocation by asking the patient to walk along a flat, hospital corridor until they need to stop due to leg pain. This will be measured at 0, 3 and 6 months.

The secondary endpoint will be through patient questionnaires and scored by an independent observer at baseline, 3 and 6 months.

Ankle-brachial pressure index will be measured by an independent vascular scientist at the start and end of the study.

Patient satisfaction will be measured at 3 months using a self-reported questionnaire.

Adherence to exercise will be measured through submission of walking logs at 1, 2 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Arterial claudication with ABPI <0.9 or post-treadmill pressure drop of >20mmHg
* Able to walk 50 metres unaided
* Willing to try and give up smoking
* Willing to take antiplatelet, rivaroxaban and statin
* Has a smartphone or pedometer or watch
* Has an email account
* Adult > 18 years old
* Able to give informed consent

Exclusion Criteria:

* Nocturnal foot pain or tissue loss
* Use of walking stick, frame or wheelchair
* Severe COPD or heart failure or arthritis
* Home oxygen
* Major amputation and non-limb wearer
* Severe hearing or visual impairment
* Prior failed exercise regime
* Prior falls
* Cognitive impairment
* Unable to work due to severity of claudication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in absolute walking distance | 3 and 6 months post randomisation
  Indoor flat surface walking distance until leg pain stops patient walking.

SECONDARY OUTCOMES:
Change in disease specific quality of life | 3 and 6 months post randomisation
  Intermittent Claudication Questionnaire (0 best - 100 worst)
Unplanned revascularisation | 6 months
  Any endovascular, open or hybrid revascularisation during follow up
Patient satisfaction | 3 months
  Patient satisfaction questionnaire (1 would never recommend - 5 would strongly recommend)
Adherence | 1, 2 and 3 months
  Adherence with 2 hours exercise per week (judged via submitted walking logs)

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Thapar, PhD, Principal Investigator — Mid and South Essex Hospitals NHS Foundation Trust
Locations (1):
- Mid and South Essex Hospitals NHS Foundation Trust, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full data set will be made available to other researchers upon publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication
Access Criteria: Upon request to PI